CLINICAL TRIAL: NCT04088123
Title: Investigation of Anti-platelet Drug Single Dose Exposure on Platelet mRNA Splicing in Healthy Subjects
Brief Title: Impact of Anti-platelet Drug Exposure on Platelet mRNA Splicing in Healthy Subjects
Status: Withdrawn | Type: Observational
Why Stopped: Inability to commence enrollment at institution, terminated on 9/23/20
Sponsor: George Washington University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Shenandoah University (Other); The GW Medical Faculty Associates (Other)
Responsible Party: Principal Investigator, Travis J. O'Brien, Associate Professor of Pharmacology and Physiology, George Washington University
Other Study IDs: NCR191544; U54MD010723 (NIH); Pharmacy Faculty Fund (Other Grant/Funding Number: Bernard J Dunn School of Pharmacy, Shenandoah University); PIND 144269 (Other: US FDA IND Exemption)
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Thrombosis; Artery
MeSH Terms: conditions — Thrombosis | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following materials will be obtained from each participant. Blood for RNA (RNAseq) and DNA (genotyping) and platelet activity analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Patients: The study design will involve analysis of platelet splicing/activity before and after exposure to a single, 180 mg loading dose of ticagrelor. All subjects will be cardiovascular healthy.
  Interventions: Drug: Ticagrelor Oral Tablet [Brilinta]

INTERVENTIONS:
Drug: Ticagrelor Oral Tablet [Brilinta] — A single loading dose of ticagrelor (180 mg) will be administered to each participant in this study.
  Other Names: Brilinta

SUMMARY:
The purpose of this pilot study is to determine how the anti-platelet drug, ticagrelor, impacts platelet mRNA splicing after a single loading dose in 10 healthy participants. These results will be valuable in that they will help inform our analysis of platelet RNA splicing after a thrombotic event.

DETAILED DESCRIPTION:
There is nothing known on how differential splicing in platelets is impacted by of P2Y12 inhibition by anti-platelet agents. Consequently, the focus of this longitudinal pilot study will be to determine the impact of a single ticagrelor loading dose (180 mg), our "model" anti-platelet drug, on platelet RNA splicing in 10 healthy individuals.

It will test the hypothesis that ticagrelor exposure does not significantly alter platelet mRNA splicing. It will involve administering a single loading dose (180 mg) of ticagrelor to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years-old
* Speak and understand English

Exclusion Criteria:

* History of blood clotting/bleeding disorders
* Current medications that are CYP3A4 inhibitors/inducers
* Current medications that their pharmacokinetics is impacted by ticagrelor (i.e. simvastatin, lovastatin, digoxin) per FDA recommendations.
* Diagnosed with arterial or venous thrombosis
* Active cancer diagnosis
* Pregnant
* Hepatic impairment including active hepatitis infection or cirrhosis
* Current hormonal contraception
* Currently taking aspirin or anti-platelet drugs. If patient has recently taken an NSAID, the last dose should have been discontinued based established criteria

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy patients who meet our inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Measurement of the Change in Platelet Activity From Baseline after Drug Administration | Comparison made 2.5 hours following drug administration
  As determined by the VerifyNow P2Y12 Assay
Measurement of the Change in Platelet mRNA splicing From Baseline after Drug Administration | Comparison made 2.5 hours following drug administration
  As determined by RNAseq analysis
Measurement of Ticagrelor Pharmacokinetics After Drug Administration | Comparison made 2.5 hours following drug administration
  Drug and its major metabolite levels will be measured by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Travis J O'Brien, PHD, Principal Investigator — George Washington University
Locations (2):
- United States (2):
  - The George Washington University School of Medicine and Health Sciences, Washington D.C., District of Columbia
  - Shenandoah University Bernard J. Dunn School of Pharmacy, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with researchers. Only aggregate data from the study